CLINICAL TRIAL: NCT02269878
Title: The Effect of FAS and FAS Ligand Genetic Polymorphisms on the Clinical Outcome of Patients With Malignant Pleural Mesothelioma Treated With Platinum-Based Regimens
Brief Title: Effect of FAS and FAS Ligand Polymorphisms on Patients With Platinum-Based -Treated Malignant Pleural Mesothelioma
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abdo Mohammed Salem, African Union organization St. Abbsia, Cairo, Egypt, Ain Shams University
Other Study IDs: Master (No14)
Record Dates: First submitted 2014-10-11; First posted 2014-10-21 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- people with MPM with Thymine/Thymine,Thymine/cytosine genotype: according to Single nucleotide polymorphism analysis of rs 763110, people have one of the following genotypes, Thymine/Thymine,Thymine/Cytosine,Cytosine/Cytosine. we will assign Thymine/Thymine, Thymine/Cytosine to group one and Cytosine/Cytosine to group two. for rs 1800682 people will have one of the following genotypes Adenine/Adenine, Adenine/Guanine or Guanine/Guanine.
- people with MPM, Cytosine/Cytosine genotype: according to Single nucleotide polymorphism analysis of rs 763110, people have one of the following genotypes, Thymine/Thymine,Thymine/Cytosine,Cytosine/Cytosine. we will assign Thymine/Thymine, Thymine/Cytosine to group one and Cytosine/Cytosine to group two. for rs 1800682 people will have one of the following genotypes Adenine/Adenine, Adenine/Guanine or Guanine/Guanine.

SUMMARY:
To Study the Effect of Polymorphisms in Fas Ligand Gene Promoter Region (rs 763110) and Fas gene (rs1800682) on Platinum-Based regimens used in treatment of malignant pleural mesothelioma (MPM)

DETAILED DESCRIPTION:
This study tries to find a correlation between single nucleotide polymorphisms (SNP) found in promoter region of Fas Ligand gene (rs 763110) and Fas (rs1800682) and clinical outcome on patients with MPM treated with platinum-Based agents as first line. the patients will have one of three following genotypes : Thymine/Thymine, Thymine/Cytosine or Cytosine/Cytosine (for Fas ligand polymorphism) and Adenine/Adenine, Adenine/Guanine or Guanine/Guanine ( for Fas polymorphism).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed Malignant Pleural Mesothelioma
* Age of 18 years or more.
* first-line chemotherapy with platinum-Based agents

Exclusion Criteria:

* history of prior malignancy.
* pregnancy or lactation or any other reason preventing him from taking platinum-Based chemotherapy (AST more than 2.5* Upper Limit of Normal or Serum bilirubin more than 1.5* Upper Limit of Normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with malignant pleural mesothelioma (MPM)
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
response rate | After 6 cycles of chemotherapy (each cycle is 21 days )
  Tumor response will be evaluated after the third (initial evaluation response) and the sixth (confirmation of initial response) chemotherapy cycle according to the modified Response Evaluation Criteria in Solid Tumors. Patients will be assigned to one of following groups: complete response (CR), Partial response (PR), Stable disease (SD) and progressive disease (PD).

SECONDARY OUTCOMES:
progression free survival (PFS) | one year
  Progression-free survival (PFS) time is defined as the time from day 1 of chemotherapy to the day of documented disease progression or to death from any cause
overall survival (OS) | one year
  time is defined as the time from day 1 of chemotherapy to death from any cause.
estimation of treatment related toxicity | during the chemotherapy period, average duration 4 months
  Hematologic (anemia, neutropenia, and thrombocytopenia) and non hematologic (nausea/vomiting, alopecia and nephrotoxicity) toxicities will be evaluated according to the National Cancer Institute-Common Toxicity Criteria. The worst degree of toxicity experienced throughout the treatment is used for the analysis. Toxicities of grade 2 or higher will be considered as clinically relevant.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasia, Egypt